CLINICAL TRIAL: NCT04724330
Title: Healthy for 2/Healthy for U: A Pragmatic Randomized Clinical Trial to Limit Gestational Weight Gain and Prevent Obesity in Johns Hopkins Prenatal Care Practices
Brief Title: Pragmatic Randomized Clinical Trial to Limit Weight Gain in Pregnancy and Prevent Obesity
Acronym: H42/H4U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00255969; R18DK122416-01A1 (NIH)
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Weight Gain; Postpartum Weight Retention; Childhood Obesity; Gestational Diabetes; Overweight and Obesity
MeSH Terms: conditions — Gestational Weight Gain; Pediatric Obesity; Diabetes, Gestational; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy for Two/Healthy for You (H42/H4U) (Experimental): Those assigned to the intervention group will receive the H42/H4U health coaching intervention during pregnancy and 12 weeks postpartum.
  Interventions: Behavioral: Healthy for Two/Healthy for You
- Usual Care Comparison Group: Maintain Health in Pregnancy (mHIP) (No Intervention): Those assigned to the Usual Care comparison group, mHIP, will receive typical, evidence- and guideline-based experience in the prenatal care clinics.

INTERVENTIONS:
Behavioral: Healthy for Two/Healthy for You — ~10 month (early pregnancy to 12 weeks postpartum), remotely-delivered, behavioral lifestyle intervention including health coach contacts (via phone, videoconference, and email/MyChart) and an interactive web-based platform.
  Other Names: H42/H4U
  Arms: Healthy for Two/Healthy for You (H42/H4U)

SUMMARY:
Healthy for Two, Healthy for You (H42/H4U) is an innovative evidence-based pregnancy/postpartum health coach intervention that is remotely-delivered (phone coaching using motivational interviewing, web-based platform, mobile phone behavioral tracking). The aim of this randomized controlled trial (RCT) is to embed H42/H4U into Johns Hopkins prenatal care clinics that serve a racially and economically diverse population, leveraging existing staff as trained health coaches to test its effectiveness and implementation. The investigators hypothesize that women in the H42/H4U arm will have lower gestational weight gain and lower rates of gestational diabetes, without an increase in low birth weight infants, and that implementation into the investigators' prenatal care clinics will be feasible and scalable.

DETAILED DESCRIPTION:
Despite two decades of public health efforts to combat obesity, rates continue to rise and racial disparities persist. There is an urgent need to re-focus obesity prevention efforts onto young adults, particularly reproductive age women. 23% of women (vs. 13% of men) gain ≥20 kg from age 18 to 55 years, with the highest weight gain in African American women who gain > 1kg/year. Importantly, weight gain of ≥20 kg is associated with development of type 2 diabetes (DM), other obesity-related comorbidities and greater mortality. For women who become pregnant, pregnancy provides an important opportunity for obesity and DM prevention, as excessive gestational weight gain (GWG) and pregnancy complications [e.g. gestational diabetes (GDM)], increase future DM risk. Promoting healthy GWG through behavioral interventions may prevent these pregnancy complications, but importantly has great potential for long-term, sustainable benefits to prevent postpartum weight retention (PPWR) and future obesity and DM, in women and the women's children.

With the publication of the LIFE-Moms consortium's results, there is now strong evidence from efficacy trials showing that limiting GWG is achievable and associated with improved exercise and dietary behaviors. Several notable research gaps and next steps have emerged from the LIFE-Moms' studies, which the investigators address in this pragmatic trial. Because these studies were designed to test the efficacy of behavioral weight management on GWG, interventions were resource intensive (i.e. in-person counseling and with limited online and mobile technologies), without a focus on program implementation and sustainability in routine prenatal care settings and lacking intervention in the vulnerable postpartum period. To address these critical evidence gaps and reduce obesity associated with the pregnancy/postpartum periods, the next step is to integrate and test an evidence-based lifestyle intervention in pregnancy and postpartum that utilizes remote delivery of counseling, enables self-monitoring by patients using mobile and online technologies and supports obstetric providers and clinics to optimize care for women at high risk for obesity and future DM.

The investigators' experienced team created and tested Healthy for Two / Healthy for You (H42/H4U). H42/H4U is an innovative evidence-based pregnancy/postpartum health coaching intervention that is remotely-delivered (phone coaching using motivational interviewing + web-based platform + mobile phone behavioral tracking). The aim of this R18 pragmatic randomized controlled trial (RCT) is to embed H42/H4U into prenatal care clinics that serve a racially and economically diverse population, leveraging existing staff as trained health coaches and community health workers (CHWs), to test its effectiveness and implementation.

The investigators hypothesize that women in the H42/H4U arm will have lower GWG and lower rates of GDM, without an increase in low birth weight infants, and that implementation into the investigators' prenatal care clinics will be feasible and scalable. The investigators will rigorously test this hypothesis through the following Specific Aims:

Aim 1. Test the effectiveness of H42/H4U integrated into prenatal care compared with Usual Care among 380 pregnant and postpartum women enrolled from 6 prenatal clinics on:

A. Primary outcome: GWG (37 week minus baseline pregnancy [≤15 week gestation] weight) B. Maternal secondary outcomes: Proportion with excessive GWG; GDM incidence; PPWR at 6 months after delivery C. Infant secondary outcomes: Weight at birth, 4 and 6 months. D. Other outcomes: Maternal health behaviors (diet, physical activity, breastfeeding); Maternal wellness (depression, sleep and stress)

Aim 2. Assess organizational factors that impact the implementation of the intervention into prenatal care clinics, including costs of intervention delivery and provider and staff satisfaction to inform future dissemination.

A. Provider and staff perspectives, including satisfaction, workflow barriers and potential for sustainability, using qualitative semi-structured interviews (n=15 at baseline and end of study).

B. Cost analysis to assess intervention delivery costs and the return on investment (ROI) of H42/H4U.

This study will advance a potentially powerful, prenatal care-based strategy to reduce obesity in young adult childbearing women and thereby the intergenerational effects on the women's children. The investigators' interdisciplinary team brings together engaged academic and community-based obstetricians, the investigators' health system's population health program and researchers with experience in developing, testing and implementing behavioral interventions in both pregnant and non-pregnant adults in real world settings to enable wide dissemination. Ultimately, the investigators' goal is to design and produce an effective and scalable behavioral strategy, integrated into clinical practice that will: 1) reduce excessive GWG and its associated pregnancy complications, 2) reduce future obesity, DM and other obesity-related complications in mothers and the mothers' children, and 3) ensure high quality care delivery that prevents obesity and DM through a population health approach to prenatal care.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18
* Singleton pregnancy
* ≤15 weeks gestation with documented prenatal weight and height in electronic health record
* Body mass index ≥ 25.0 kg/m2
* English-speaking
* Has smartphone, laptop or tablet and willing to use it for this study
* Has email address and willing to use for this study

Exclusion Criteria:

* BMI <25 kg/m2
* Multiple fetuses
* History of pre-gestational Type 1 or Type 2 diabetes or taking diabetes medication for treatment of diabetes prior to first prenatal visit
* Prior history of severe preeclampsia, pre-term birth (< 32 weeks gestation)
* Poorly controlled blood pressure (> 160/100 mmHg)
* Substance use disorder or positive urine toxicology (except for THC) for illicit substances (screening done as part of routine care)
* Psychiatric hospitalization in last 12 months or diagnosis of severe mental illness that is not well controlled
* Active diagnosis of an eating disorder
* Unable to walk 1 block without pain or shortness of breath
* No email address
* Unable to speak or read in English
* Planning to move in next 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Total gestational weight gain | At 37 weeks in pregnancy
  Difference between weight (lbs) at 37 weeks and baseline first trimester weight, measured prior to 15 weeks gestation.

SECONDARY OUTCOMES:
Number of participants who gained excess weight | At 37 weeks in pregnancy
  Number of participants who gained above the Institute of Medicine recommended weight gain goal.
Incidence of gestational diabetes mellitus | At 37 weeks in pregnancy
  Defined and validated by electronic health record diagnosis.
Postpartum weight retention | 6 months after delivery
  Difference between baseline (≤ 15 weeks gestation weight) and 6 month post delivery maternal weight (lbs).
Infant weight | At 6 months of age
  Weight (lbs) of infant assessed by electronic health record.
Proportion of low birth weight infants | At time of birth/delivery
  Proportion of infants weighing < 2500 grams at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Bennett, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Health System and University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drabo EF, McKinney CD, Martin LM, Nair D, Coughlin JW, Chen T, Borahay MA, Wang NY, Bennett WL. Protocol for the economic evaluation of the "Healthy for Two/Healthy for You" pragmatic lifestyle intervention in prenatal care to reduce gestational weight gain and gestational diabetes mellitus. Contemp Clin Trials. 2025 Sep;156:108037. doi: 10.1016/j.cct.2025.108037. Epub 2025 Jul 31. PMID 40752820
- [Result] Bennett WL, Coughlin JW, Henderson J, Martin S, Yazdy GM, Drabo EF, Showell NN, McKinney C, Martin L, Dalcin A, Sanders R, Wang NY. Healthy for Two/Healthy for You: Design and methods for a pragmatic randomized clinical trial to limit gestational weight gain and prevent obesity in the prenatal care setting. Contemp Clin Trials. 2022 Feb;113:106647. doi: 10.1016/j.cct.2021.106647. Epub 2021 Dec 8. PMID 34896296